CLINICAL TRIAL: NCT00799435
Title: Treatment With Glucagon-Like Peptide-1 Receptor, Exenatide, in Patients With Diabetes and Heart Failure With Normal Left Ventricular Ejection Fraction
Brief Title: Evaluating the Use of Exenatide in People With Type 2 Diabetes and Diastolic Heart Failure
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit adequate Sample Size who met the entry criteria
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Aguilar, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 613; 1K01HL092585 (NIH); 1K01HL092585-01 (NIH); H-22906 (Other: Baylor College of Medicine)
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure, Diastolic
Keywords: Diabetes; Diastolic Heart Failure; Aortic Stiffness; Exenatide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure, Diastolic; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Participants will receive usual care for 12 weeks. The care will be dictated by the primary physician and/or diabetologist caring for the participant. Efforts will be made to ensure that all participants receive standard measures as indicated by guidelines, with a particular emphasis on blood pressure control and glucose control.
- 2 (Experimental): Participants will receive exenatide for 12 weeks.
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — 5 μg of exenatide subcutaneously twice a day for 4 weeks, followed by 10 μg of exenatide subcutaneously twice a day for an additional 8 weeks
  Other Names: Byetta
  Arms: 2

SUMMARY:
People with type 2 diabetes experience heart failure more often than do people without diabetes. This may be due to increased stiffness in the heart as a result of diabetes. This study will examine whether exenatide, a medication used to treat diabetes, may have beneficial effects on the heart in people with type 2 diabetes and heart failure.

DETAILED DESCRIPTION:
Diastolic heart failure is a life-threatening condition that occurs when the ventricles of the heart become stiff and do not fully relax, preventing the heart from properly filling with blood. The circulation of blood then backs up, and blood collects in the body's organs, primarily the lungs. However, people with diastolic heart failure may have a normal ejection fraction, which is a measure of the amount of blood that the heart pumps out with each heart beat. Having type 2 diabetes may increase the risk of diastolic heart failure. Also, people with both heart failure and type 2 diabetes are more likely to experience poor health and even death than are people with only heart failure. It is possible that diabetes leads to increased stiffness of the ventricles and the aorta, which is the main blood vessel into which the heart empties. Exenatide, part of a class of medications known as glucagon-like peptide-1 (GLP-1) receptor agonists, is a new medication that is currently used to treat elevated blood sugar levels in people with diabetes. Some studies have shown that this class of medications may have a positive effect on the heart and blood vessels. The purpose of this study is to determine the effect that exenatide has on aortic and left ventricular stiffness in people who have type 2 diabetes and diastolic heart failure.

This 12-week study will enroll adults with type 2 diabetes and diastolic heart failure with normal ejection fraction. At a baseline study visit, participants will undergo a physical examination, blood pressure and heart rate measurements, a blood collection, an echocardiogram to obtain images of the heart, and a non-invasive test that measures blood flow in the aorta. Participants will then be randomly assigned to receive either exenatide or usual care. Participants who receive exenatide will inject the medicine twice a day for 12 weeks. At Week 4, these participants will attend a study visit to adjust the medication dosage and to report any problems, and at Week 6, study staff will follow up with participants by phone. All participants will attend a study visit at Week 12 for repeat baseline testing.

ELIGIBILITY:
Inclusion Criteria:

* Stable New York Heart Association (NYHA) Class II-IV heart failure symptoms for at least 4 weeks before study entry
* Diagnosis of diastolic heart failure with a normal ejection fraction
* Admitted to the hospital with a diagnosis of heart failure in the 12 months before study entry
* Type 2 diabetes

Exclusion Criteria:

* Unstable angina, heart attack, coronary artery bypass surgery, or angioplasty in the 3 months before study entry
* Angina with exertion
* Technically inadequate echocardiogram
* Atrial fibrillation or atrial flutter
* Severe valvular heart disease
* Significant kidney insufficiency (serum creatinine greater than 2.0 mg/dL or require hemodialysis)
* Conditions that may be associated with changes in markers of fibrosis or collagen turnover (e.g., ongoing or active rheumatological disease, requiring significant anti-inflammatory agents, immunosuppression, pulmonary fibrosis, active cancer)
* Significant history of active substance abuse
* Type 1 diabetes
* Type 2 diabetes requiring chronic insulin use before study entry
* Active thiazolidinedione (TZD) use, because TZDs have been shown to worsen volume retention and may exacerbate signs and/or symptoms of heart failure
* Pregnant or breastfeeding
* Hypertrophic cardiomyopathy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Aguilar, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Participants will receive usual care for 12 weeks. The care will be dictated by the primary physician and/or diabetologist caring for the participant. Efforts will be made to ensure that all participants receive standard measures as indicated by guidelines, with a particular emphasis on blood pressure control and glucose control.
- Exenatide Group: Participants will receive exenatide for 12 weeks.
  Exenatide: 5 μg of exenatide subcutaneously twice a day for 4 weeks, followed by 10 μg of exenatide subcutaneously twice a day for an additional 8 weeks
Period: Overall Study
Arm/Group | Control Group | Exenatide Group
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Participants will receive usual care for 12 weeks. The care will be dictated by the primary physician and/or diabetologist caring for the participant. Efforts will be made to ensure that all participants receive standard measures as indicated by guidelines, with a particular emphasis on blood pressure control and glucose control.
- Exenatide: Participants will receive exenatide for 12 weeks.
  Exenatide: 5 μg of exenatide subcutaneously twice a day for 4 weeks, followed by 10 μg of exenatide subcutaneously twice a day for an additional 8 weeks
- Total: Total of all reporting groups
Arm/Group | Usual Care | Exenatide | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — texas
  Participants
    United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Aortic Stiffness, as Measured by the Change in the Mean Aortic Pulse Wave Velocity
Time Frame: Measured at Week 12
Population: For the usual care, data were obtained for only person, but data was collected only at baseline and follow-up data were not collected. For the exenatide arm, data were collected for only one participant at baseline and follow-up.
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | Usual Care | Exenatide
Number analyzed (Participants) | 1 | 1
m/sec
  Baseline Pulse Wave Velocity | 11.4 (0) | 9.3 (0)
  Follow-up Pulse Wave Velocity | NA (NA) — Could not obtain technically obtain an adequate follow-up PWV reading | 10.2 (0)

2. Secondary Outcome: Changes in Left Ventricular Diastolic Stiffness, Serum Levels of Advanced Glycation End Products, Serum Biomarkers of Collagen Synthesis, and Serum Levels of Brain Natriuretic Peptide
Description: Given the cessation of trials, the biomarkers analyses and diastolic function measures were not performed.
Time Frame: Measured at Week 12
Population: Given the cessation of trials, the biomarkers analyses and diastolic function measures were not performed.
Arm/Group | Usual Care | Exenatide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Standard Care: Participants will receive usual care for 12 weeks. The care will be dictated by the primary physician and/or diabetologist caring for the participant. Efforts will be made to ensure that all participants receive standard measures as indicated by guidelines, with a particular emphasis on blood pressure control and glucose control.
Arm/Group | Standard Care | Exenatide
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
The study was stopped due to difficulties enrolling and fulfilling entry criteria

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No